CLINICAL TRIAL: NCT05852457
Title: Prospective Evaluation of the Clinical Utility of Endoscopic Closure Using a Dual Action Tissue (DAT) Clip
Brief Title: Evaluation of the Clinical Utility of Endoscopic Closure Using a Dual Action Tissue (DAT) Clip
Status: Recruiting | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1931144
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-01

CONDITIONS: GI Bleeding; Perforation Colon; Perforation Bowel; Perforation Duodenal; Perforated Bowel; Fistula
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Intestinal Perforation; Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: DAT Clip — All patients scheduled to undergo endoscopic procedures as medically indicated will be considered for the study. Data will be prospectively recorded according to the data collection form. The use of the DAT clip will be performed as medically indicated and consistent with the indications for endoscopic clipping (e.g., management of bleeding, treatment of fistulas, perforations, tissue approximation). The investigators on this project will also oversee the medical care of all patients that will participate in the study. Therefore, follow-up will be carried out as medically indicated and no clinical visits will be needed specifically for the purpose of this study.

SUMMARY:
This study is designed as a multicenter prospective data recording study to document the performance of the DAT clip as part of standard medical care of patients. No experimental interventions will be performed.

DETAILED DESCRIPTION:
Endoscopic clipping devices are instruments designed to achieve tissue approximation during gastrointestinal endoscopy. Although endoscopic clips were initially developed for the primary purposes of accomplishing hemostasis of focal gastrointestinal bleeding, the indications for endoscopic clipping have expanded to include closure of perforations and fistulas, securing positioning of catheters and stents as well as to provide a radio-opaque markers to direct endoscopic, radiological, and surgical therapy.

Traditionally, through-the-scope (TTS) clipping devices consist of 2 main components: metallic double pronged clips and delivery/deployment catheter-handle assembly. TTS clips are the most used devices for both hemostasis and defect closure given the familiarity and ease of use. However, larger defects or those in a difficult position within the GI tract can be difficult to close using conventional TTS clips alone, given the inherent restrictions in clip opening width and inability to approximate large gaps firmly and securely. Incomplete closure can have serious consequences, including delayed bleeding and need for additional interventions including surgery for treatment of acute perforations.

The Dual Action Tissue (DAT) clip is a novel, Federal Drug and Administration (FDA) approved commercially available 3-arm TTS clip designed for endoscopic closure of large defects. Compared to conventional TTS clips, the DAT clip has an additional center post or fixed column in the middle position. The two arms of the DAT clip operate independent of each other, with an overall maximum opening width angle of 60 degrees. Opening and closing of each arm is controlled by two color-coded handles, which facilitates distinguishment of the clip arms during operation. The arm on one side of the DAT clip is opened to clamp the edge of a defect. The clamped mucosa can then be pulled close to the other side of the defect. The second arm of the DAT is then opened to clamp the opposite edge. Once both edges of the defect are secured by the arms of the DAT clip, the clip can then be deployed by firmly pressing and releasing both handles simultaneously.

Experimental studies using the DAT clip have confirmed its safety and efficacy and shown it to be easy to operate, safe and effective for defect closure. Our initial experience in 6 cases (unpublished data) supports its safety and its utility as an additional endoscopic tool in our armamentarium for challenging tissue approximation. However, more data is needed to evaluate the performance and the role of the DAT clip. The purpose of this study is to prospectively evaluate our experience with the DAT clip as part of routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients scheduled to undergo endoscopic procedures as part of their routine care in which endoscopic clip closure is clinically indicated:

Treatment of bleeding Treatment of perforation and/or fistulas Tissue approximation for mucosal gaps associated with endoscopic resection (e.g., endoscopic mucosal resection, endoscopic submucosal dissection) or third space endoscopy (e.g., peroral endoscopic myotomy in the gastrointestinal tract)

Exclusion Criteria:

* Any contraindications to performing endoscopy.
* Participants in another research protocol that could interfere or influence the outcomes measures of the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled to undergo endoscopic procedures at participating centers as medically indicated will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Complete closure rate. | 12 months
  Cases in which complete tissue approximation is achieved with the use of the DAT clip- no substantial gaps are visible in the closure line.

SECONDARY OUTCOMES:
Rate of Achievement of intended targeted therapy. | 12 months
  Defined as cases in which utilization of the DAT clip accomplished the intended treatment effect (e.g., hemostasis, perforation closure)
Procedural time. | 12 months
  Measure of procedural time associated with the operation of the DAT clip for its intended purpose.
Adverse Events | 12 months
  Measured based on the rate of adverse events with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yang, MD, Principal Investigator — AdventHealth
Locations (2):
- United States (2):
  - AdventHealth Orlando, Orlando, Florida
  - Parkview Health, Fort Wayne, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Technology Assessment Committee; Chuttani R, Barkun A, Carpenter S, Chotiprasidhi P, Ginsberg GG, Hussain N, Liu J, Silverman W, Taitelbaum G, Petersen B. Endoscopic clip application devices. Gastrointest Endosc. 2006 May;63(6):746-50. doi: 10.1016/j.gie.2006.02.042. No abstract available. PMID 16650531
- [Background] Wang TJ, Aihara H, Thompson AC, Schulman AR, Thompson CC, Ryou M. Choosing the right through-the-scope clip: a rigorous comparison of rotatability, whip, open/close precision, and closure strength (with videos). Gastrointest Endosc. 2019 Jan;89(1):77-86.e1. doi: 10.1016/j.gie.2018.07.025. Epub 2018 Jul 27. PMID 30056253
- [Background] Zhang Q, Jin HY, Shen ZH, Ma XJ, Li CQ, Tang Z, Bai Y, Wang Z. Novel through-the-scope twin clip for the closure of GI wounds: the first experimental survival study in pigs (with videos). Gastrointest Endosc. 2021 Oct;94(4):850-858.e2. doi: 10.1016/j.gie.2021.04.027. Epub 2021 May 7. PMID 33965383
- [Derived] Mohammed A, Gonzaga ER, Hasan MK, Saeed A, Friedland S, Bilal M, Sharma N, Jawaid S, Othman M, Khalaf MA, Hwang JH, Viana A, Singh S, Hayat M, Cosgrove ND, Jain D, Arain MA, Kadkhodayan KS, Yang D. Low delayed bleeding and high complete closure rate of mucosal defects with the novel through-the-scope dual-action tissue clip after endoscopic resection of large nonpedunculated colorectal lesions (with video). Gastrointest Endosc. 2024 Jan;99(1):83-90.e1. doi: 10.1016/j.gie.2023.07.025. Epub 2023 Jul 21. PMID 37481003